CLINICAL TRIAL: NCT00784212
Title: A Multicenter, Single-blind, Within-subject, Placebo-controlled Proof of Concept Study to Assess the Effect of Single Oral Doses of BGG492 on the Photoparoxysmal EEG Response in Patients With Photosensitive Epilepsy
Brief Title: Effect of BGG492 on EEG in Patients With Photosensitive Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBGG492A2203; 2007-005418-38 (EudraCT Number)
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Photosensitive Epilepsy
Keywords: Photosensitive Epilepsy, photic stimulation, electroencephalogram
MeSH Terms: conditions — Epilepsy, Reflex | interventions — selurampanel

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Drug: BGG492
- Cohort II (Experimental)
  Interventions: Drug: BGG492
- Cohort III (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGG492
  Arms: Cohort 1
Drug: BGG492
  Arms: Cohort II
Drug: Placebo
  Arms: Cohort III

SUMMARY:
This study will evaluate the efficacy of BGG492 in reducing the sensitivity to flashing lights of patients with photosensitive epilepsy, using EEG as a readout.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of photosensitive epilepsy

Exclusion Criteria:

- inconsistent photoparoxysmal response when stimulated by photic stimulation

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: Photoparoxysmal response (PPR) and standardized photoparoxysmal response (SPR) determined by EEG on all treatment days. | Days 1, 2 and 3

SECONDARY OUTCOMES:
Outcome Measure: Safety and tolerability of BGG492 in patients with photosensitive epilepsy | From Day 1 until Day 33 after treatment start.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis Investigator Site
Locations (4):
- Germany (4):
  - Novartis Investigator Site, Bielefeld
  - Novartis Investigator Site, Kehl-Kork
  - Novartis Investigator Site, Kiel
  - Novartis Investigator Site, Radeberg

REFERENCES:
- [Derived] Kasteleijn-Nolst Trenite D, Brandt C, Mayer T, Rosenow F, Schmidt B, Steinhoff BJ, Gardin A, Imbert G, Johns D, Sagkriotis A, Kucher K. Dose-dependent suppression of human photoparoxysmal response with the competitive AMPA/kainate receptor antagonist BGG492: Clear PK/PD relationship. Epilepsia. 2015 Jun;56(6):924-32. doi: 10.1111/epi.13008. Epub 2015 May 11. PMID 25963722